CLINICAL TRIAL: NCT05346926
Title: Overnight and In-house 3D-printed Patient-specific Casts for Non-operative Treatment of Distal Radius Fractures - a Prospective Randomized Trial
Brief Title: Overnight and In-house 3D-printed Patient-specific Casts for Non-operative Treatment of Distal Radius Fractures
Acronym: 3D-cast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alissa Gubeli (Other)
Collaborators: Spentys (Industry)
Responsible Party: Sponsor-Investigator, Alissa Gubeli, Junior Consultant Hand Surgery, Kantonsspital Baselland Bruderholz
Organization: Kantonsspital Baselland Bruderholz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01644
Record Dates: First submitted 2022-04-17; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Radius Fracture Distal
Keywords: Distal Radius Fracture, 3D-Printing
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-printed cast (Experimental): Treatment of distal radius fracture with 3D-printed forearm cast.
  Interventions: Device: 3D-printed cast
- Conventional cast (Active Comparator): Treatment of distal radius fracture with conventional plaster cast.
  Interventions: Device: Conventional cast

INTERVENTIONS:
Device: 3D-printed cast — The 3D-printed casts are produced using 3D print technology based on software by Belgian software company: The patient's forearm is scanned with a tablet (duration: approx. 5 min), whereupon the cast is printed overnight according to the scan (duration: approx. 4h) and adjusted to the patient during the next appointment.
  Arms: 3D-printed cast
Device: Conventional cast — A conventional plaster cast is applied for treatment of the distal radius fracture.
  Arms: Conventional cast

SUMMARY:
The aim of this prospective randomized trial is the acquisition and evaluation of data to assess the relevance, feasibility and safety of forearm casts based on 3D-printing technology in the nonoperative treatment of distal radius fractures.

DETAILED DESCRIPTION:
The study design is planned according to similar studies investigating the treatment of distal radius fractures.

Upon the patient's arrival at the emergency unit, the distal radius fracture is examined following the same scheme as before. The wrist is x-rayed in two planes. If there is a distal radius fracture and none of the exclusion criteria apply, the patient is included in the study after giving their consent in writing. The patients are then assigned to the "conventional cast" group (Group A) or the "3D print cast" group (Group B) in randomized trial, either immediately during the emergency consultation or within a week during hand surgery consultation hours. For initial immobilization, a thermoplastic cast splint is used as before. Depending on the randomization, the cast is changed to a Scotchcast cast (Group A) or a 3D printed cast (Group B). Further treatment of both groups occurs based on the same algorithm as before (see below).

The cast for Group B are produced using 3D print technology based on software by a Belgian company, our collaborators: The patient's forearm is scanned with a tablet (duration: approx. 5 min), whereupon the cast is printed overnight according to the scan (duration: approx. 4h) and adjusted to the patient during the next appointment.

The patients are examined after 1, 6, 12, 26 and 52 weeks in the outpatient clinic. Follow up x rays, patient satisfaction and clinical efficacy questionnaires and clinical examinations are conducted.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Undisplaced or minimally displace distal radius fractures

Exclusion Criteria:

1. Age < 18yrs.
2. Dorsal dislocation (dp angle) >20°
3. Palmar dislocation
4. Ad latus dislocation
5. Radio-/ulnar angulation in the coronary plane
6. Symptoms of neurologic affection (Median nerve)
7. Bilateral fractures
8. Previous ipsilateral distal radius fracture
9. The patient is unable to give informed consent due to physical or mental impairment
10. The patient is unavailable for follow-up examinations (foreign country, Polytrauma, etc)
11. The patient is under legal custodianship
12. C2- or Drug-abuse or expected incompliance
13. Hypersensitivity/Allergy to one or more components of the used casts
14. Pregnancy/Intention to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Score of modified patient satisfaction questionnaire | 1 year
  quantified with questionnaire (0-12, 0=worst result)
Score of clinical effectiveness questionnaire | 1 year
  quantified with questionnaire (0-12, 0=worst result)

SECONDARY OUTCOMES:
Fracture healing | 1 year
  assessed with X-ray pictures taken during the follow-up, consolidation signs
Score on Visual Analogue Pain Scale | 1 year
  assessed using the Visual Analogue Pain Scale (0-10, 0=best result, no pain)
Amount of range of motion in degrees | 1 year
  assessed/measured by the physician with a goniometer (°, 0-360°)
Amount of grip strength in (N/kg) | 1 year
  assessed with a dynamometer (N/kg, the lower the weaker)
Score of Disabilities of Arm, Shoulder and Hand | 1 year
  assessed with Disabilities of Arm, Shoulder and Hand score (0-100, 0=best result, no impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Honigmann, PD Dr. med., Study Director — Cantonal Hosptal, Baselland
Locations (1):
- Kantonsspital Baselland, Bruderholz, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No